CLINICAL TRIAL: NCT06981702
Title: Effects of Exercıse on Chronotype, Sleep Qualıty and Depressıonal Symptom Level in Unıversıty Students Who Exercıse Regularly
Brief Title: Effects of Exercıse on Chronotype, Sleep Qualıty and Depressıon Symptom Level in Unıversıty Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nazan Ozturk, Principal Investigator, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NzOzturk
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-05

CONDITIONS: Depression, Anxiety; Chronotype; Physical Activity
Keywords: physical activity; depression; chronotype
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Active Comparator): . In our study, demographic information (age, gender, height, weight, education, marital status, occupation, where and with whom they live), additional diseases, medications used, whether they live in a rural or urban area, whether they have had any sleep problems before, and whether they have had any psychiatric diagnoses before will be recorded for all subjects. Before the exercise, students will fill out the Pittsburgh Sleep Quality Index to determine their sleep quality, the Morningness-Eveningness Scale to assess their chronotype, and the Beck Depression Inventory to measure their depressive symptom levels, and the results will be recorded. Students taking the body mechanics course will be asked to do aerobic exercises they learned in class, three days a week, including warm-up and cool-down, for a total of 60 minutes of exercise. The exercises will be performed on the same days and times each week. All exercises performed by the students for 8 weeks will be monitored by the rese
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — . In our study, demographic information (age, gender, height, weight, education, marital status, occupation, where and with whom they live), additional diseases, medications used, whether they live in a rural or urban area, whether they have had any sleep problems before, and whether they have had any psychiatric diagnoses before will be recorded for all subjects. Before the exercise, students will fill out the Pittsburgh Sleep Quality Index to determine their sleep quality, the Morningness-Eveningness Scale to assess their chronotype, and the Beck Depression Inventory to measure their depressive symptom levels, and the results will be recorded. Students taking the body mechanics course will be asked to do aerobic exercises they learned in class, three days a week, including warm-up and cool-down, for a total of 60 minutes of exercise. The exercises will be performed on the same days and times each week. All exercises performed by the students for 8 weeks will be monitored by the resea

SUMMARY:
The aimed this study is to determine the effect of regular exercise program on mood, chronotype and sleep quality in university students.

DETAILED DESCRIPTION:
The study is a quasi-experimental study with a pretest-posttest design. Demographic information (age, gender, height, weight, education, marital status, occupation, where and with whom they live), additional diseases, medications used, whether they live in a rural or urban area, whether they have had any previous sleep problems, and whether they have had any previous psychiatric diagnoses will be recorded for all subjects in the study. Before the exercise, students will fill out the Pittsburgh Sleep Quality Index to determine their sleep quality, the Morningness-Eveningness Scale to assess their chronotype, and the Beck Depression Inventory to measure their depressive symptom levels, and the results will be recorded. All exercises performed by the students for 8 weeks will be monitored by the researcher physiotherapist through weekly short individual or group interviews with the students. At the end of the eighth week, students will fill out the Pittsburgh Sleep Quality Index, Morningness-Eveningness Scale, and the Beck Depression Inventory again, and the results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Studying at Aydın Adnan Menderes University Söke Health Services College,
* Taking the body mechanics course,
* Being between the ages of 18-49,
* Being able to read, speak and understand Turkish.

Exclusion Criteria:

* Having received physical therapy services due to musculoskeletal diseases in the last 3 months,
* Having musculoskeletal diseases such as ankylosing spondylitis, chronic or structural joint diseases,
* Having congenital malpositions of the musculoskeletal system,
* Having a physical disability,
* Having undergone artificial joint replacement,
* Having multiple sclerosis, myodystrophic or other neurodegenerative diseases, Having serious diseases such as acute herniated disc, Using muscle relaxants or other drugs that affect muscle elasticity, Having a cardiovascular disease, Having a history of previous back surgery, Having a traffic accident in the last 6 months, Not being within the age range determined for the study, Having a mental disability that prevents answering the comprehension and evaluation forms.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | immediately after application
  This index includes 19 items designed to evaluate sleep quality in the last month. Subjective sleep quality consists of sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleeping pill use and daytime sleep dysfunction. Each component is evaluated on a 0-3 scale. The total score has a value between 0-21. A high total score indicates poor sleep quality. A total PSQI score greater than 5 is an indicator of a significant level of sleep disturbance. The validity and reliability studies of this scale for our country were conducted by Ağargün et al. in 1996.
Morningness-Eveningness Questionnaire - MEQ | immediately after application
  This scale helps determine when individuals are more active and awake in accordance with their biological clocks. The scale consists of a total of 19 items and includes questions aimed at determining whether individuals are morning type, evening type, or intermediate type. These questions cover topics such as individuals' sleep and wakefulness habits, performance levels in the morning and evening hours, and when they feel more energetic. The sum of the scores given to each item determines the person's morning or evening tendency: Morning individuals are more energetic in the early hours and work more efficiently in the morning. Evening individuals are more energetic in the late hours and work more efficiently in the evening. Intermediate individuals, on the other hand, can perform in a balanced manner at different times of the day without showing a clear morning or evening tendency. The total score helps classify the individual as being in accordance with their circadian rhythm. The v
Beck Depression Inventory- BDI | immediately after application
  This scale is widely used in the evaluation of depression, especially in psychiatric practices and clinical research. The BDI consists of a total of 21 items, and each item includes the basic symptoms of depression (e.g. sadness, hopelessness, sleep disorders, appetite changes, feelings of worthlessness). Each item is scored between 0 and 3. Scores increase according to the severity of the individual's symptoms, and the total score varies between 0 and 63. Individuals who score between 0 and 13 have no or mild depression. Scores between 14 and 28 indicate moderate depression. Scores between 29 and 63 indicate severe depression. A high total score indicates more severe depression. The BDI is frequently used to better understand individuals' depression levels and to monitor progress in the treatment process. The validity and reliability studies of this scale were conducted by Hisli in 1986.

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Demir Yazıcı, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydin Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No